CLINICAL TRIAL: NCT06046313
Title: A Multi-center Prospective Single Arm Clinical Study of Prolonged Ultra Low-dose Decitabine Combined With Venetoclax (Bcl-2 Inhibitor) as First Line Treatment for Elderly Acute Myeloid Leukemia and High-risk Myelodysplastic Syndromes
Brief Title: Prolonged Ultra Low-dose Decitabine Plus Venetoclax for Primary Diagnosed Elderly AMLK/MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Weiyan Zheng, Clinical Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT202300032C
Record Dates: First submitted 2023-04-13; First posted 2023-09-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Acute Myeloid Leukemia Myelodysplastic Syndrome
  Interventions: Drug: Decitabine for Injection; Drug: VENCLYXTO

INTERVENTIONS:
Drug: Decitabine for Injection — 6mg/m2, ivgtt qd d1-10
  Other Names: Dacogen; 5-Aza-29-deoxycytidine
Drug: VENCLYXTO — 100mg p.o.d1, 200mg p.o.d2, 400mg p.o.d3-21,adjust by blood concentration
  Other Names: VENLEXTA

SUMMARY:
To explore the efficacy and safety of prolonged low-dose decitabine (10 days of 6mg/m2) plus venetoclax (3 weeks/cycle) regimen in primary diagnosed elderly or frail AML/ high-risk MDS.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) are hematological malignancies. Some patients are over 65 years old, have poor response to traditional chemotherapy, and rarely have the opportunity to receive allogeneic hematopoietic stem cell transplantation, resulting in poor prognosis and short survival.

In recent years, with the advent of molecular targeted drugs Bcl-2 inhibitors, the treatment of elderly AML/ high-risk MDS has achieved breakthrough progress. In particular, the combination of demethylated drugs (decitabine/azacidacidin) and Bcl-2 inhibitors of chemotherapy-free regimen has been recommended by NCCN as the first-line treatment for elderly and frail patients.

However, how to achieve the optimal combination of decitabine and Bcl-2 inhibitors is an urgent problem to be solved.

Our previous pilot trial showed that prolonged low-dose decitabine combined with venetoclax (Bcl-2 inhibitor) resulted in higher complete remission rate, longer disease-free survival, and lower treatment-related risks.

The purpose of this study was to expand the multi-center sample to explore the efficacy and safety of prolonged low-dose decitabine plus venetoclax regimen in primary diagnosed elderly or frail AML/ high-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with acute myeloid leukemia (non-acute promyelocytic leukemia)/high-risk myelodysplastic syndrome before admission.

   Diagnostic criteria refer to 2016 WHO classification.
2. Age 60 or older.
3. The scores of physical fitness in the Eastern Tumor Cooperative group (ECOG) ranged from 0 to 3(see Appendix 1).
4. Creatinine clearance ≥30 mL/min(as assessed by the Cockcrod-Gault formula [Cockcroft et al 1976] [13] or the estimated glomerular filtration rate [eGFR] from the Kidney Drink adjustment formula .
5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤3× upper limit of normal range (ULN), total bilirubin ≤2×ULN.
6. Echocardiography (ECHO) showed left ventricular ejection fraction (LVEF)≥50% (AHA 2016).
7. Life expectancy >8 weeks.
8. Sign the informed consent voluntarily, and understand and comply with the requirements of the study.

Exclusion Criteria:

1. Age <60 years old.
2. Treated patients who had received various chemotherapy regiments.
3. Present clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional scale (see Appendix 2), or history of myocardial infarction in the 6 months prior to screening.
4. Other serious diseases that may limit participation in the trial (e.g. advanced infections, uncontrolled diabetes).
5. Those who cannot understand and follow the research plan or sign the informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CR+CRi) | at Week 8
  Assessment of CR(CR=CR+CRi) at Week 8

SECONDARY OUTCOMES:
MRD | at Week 8
  Assessment of minimal residual disease (MRD) at Week 8
EFS | up to 2 years after induction therpy
  Evaluation of Event-free survival (EFS)
OS | up to 2 years after induction therpy
  Evaluation of overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Weiyan Zheng, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China